CLINICAL TRIAL: NCT01642446
Title: A Randomized Control Clinical Trial Between Precise Hepatectomy and Combined Interventional Treatment on Hepatocellular Carcinoma (HCC) With Cirrhotic Portal Hypertension
Brief Title: Optimal Treatment on Hepatocellular Carcinoma (HCC) With Cirrhotic Portal Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yunfei Yuan, Prof., Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20125010Y
Record Dates: First submitted 2012-07-12; First posted 2012-07-17 (Estimated); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: Hepatocellular Carcinoma(HCC); Cirrhotic Portal Hypertension
Keywords: precise hepatectomy; hepatocellular carcinoma; cirrhotic; portal hypertension; safety; combined interventional treatment
MeSH Terms: conditions — Carcinoma, Hepatocellular; Hypertension, Portal

STUDY DESIGN:
Intervention Model Description: transartery embolization chemotherapy, infusion of Chemoembolization was performed using 30 mg/m2 of epirubicin, 200 mg/m2 of carboplatin, and 4mg/m2 of mitomycin C (MMC), mixed with 2-5 mL lipiodol. Then up to 20 mL of additional pure lipiodol was injected into the tumor-feeding artery until stasis of blood flow in the target artery was observed
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- surgery (Experimental): Precise hepatectomy
  Interventions: Procedure: Precise hepatectomy
- combined intervention (Active Comparator): transcatheter hepatic arterial chemoembolization and/or ablation
  Interventions: Other: Combined intervention (chemoembolization/ablation)

INTERVENTIONS:
Procedure: Precise hepatectomy — Precise hepatectomy
  Arms: surgery
Other: Combined intervention (chemoembolization/ablation) — transcatheter hepatic arterial chemoembolization and/or ablation
  Arms: combined intervention

SUMMARY:
There is no consensus about the optimal treatment of hepatocellular carcinoma (HCC) with cirrhotic portal hypertension, While this group of patients are classified as hepatectomy contraindication according to guidelines from National Comprehensive Cancer Network (NCCN) and American Association for the Study of Liver Diseases (AASLD). With improvement of surgical technique, preoperative evaluation, and perioperative management,especially the Precise Hepatectomy Technique, more and more studies confirmed the safety of surgical intervention to hepatocellular carcinoma (HCC) patients with cirrhotic portal hypertension.However, most of the previous studies were either retrospective or with small samples.

The investigators project is a prospective randomized controlled trial, planning to compare the safety, efficacy and quality of life between precise hepatectomy and combined interventional treatment on hepatocellular carcinoma (HCC) with cirrhotic portal hypertension, to make a further understanding of optimal strategy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of hepatocellular carcinoma patients, in accordance with HCC Professional Committee of the Chinese Anti-Cancer Association 2001 "Clinical Diagnosis of Primary Liver Cancer and Staging Criteria"
* solitary tumor ≤5cm, or three or fewer lesions none ≤3cm，As Milan criteria
* History of hepatitis B or HBsAg positive
* Cirrhosis and portal hypertension
* No treatment on liver cancer before
* KPS score ≥ 70
* The age of 18 to 65 years
* Child-Pugh A or B (Class B, scoring no more than 7 points)
* Baseline laboratory test comply with the following criteria:

  * White blood cell ≥ 1.0×109/L
  * Platelet ≥ 25×109/L
  * Hemoglobin ≥ 80g/L
  * Serum ALT,AST ≤ 3×upper limit of normal (ULN)
  * Serum creatinine ≤ 1.5 × ULN
  * INR<1.5, or prothrombin time <ULN +4 sec
  * Albumin ≥30g/L
  * Total bilirubin ≤34mmol/L
* Informed consent with signature and time
* Good patient compliance
* The surgical group patients received radical hepatectomy. Radical surgery is defined as: complete resection of visible tumor, R0 resection margins, and also including:

  * The number of tumors is less than 3
  * No tumor thrombus found in major branch of the portal veins, hepatics, inferior vena cava or bile duct
  * No hepatic hilar lymph node metastasis
  * No extrahepatic metastasis

Exclusion Criteria:

* extrahepatic metastasis; With metastasis in major branch of portal vein, hepatic vein
* History of hepatitis C or HCV-Ab positive
* Pugh Child-Pugh C, or with massive ascites or had a history of hepatic encephalopathy, or Upper digestive tract bleeding
* Poor physical condition or cachexia
* During the past 12 months just before the study, there had been any of the following: myocardial infarction, severe/unstable angina, coronary artery bypass graft surgery, congestive heart failure, cerebrovascular accident (including transient ischemic attack), pulmonary embolism; arrhythmia according to the NCI-CTCAE ≥ grade 2, QTc interval extension (male> 450 ms, female> 470 ms);
* Renal insufficiency, need peritoneal dialysis or hemodialysis
* Serious dysfunction of other organs
* History of second primary malignant tumors
* Known or new evidence of brain or leptomeningeal disease
* Hemophilia or bleeding tendency, and are taking therapeutic doses of coumarin derivative anticoagulant therapy drugs
* Pregnant or lactation, all female patients with childbearing potential must have a pregnancy test (serum or urine) within 7 days after enrollment,and the result is negative
* History of organ transplantation
* Known HIV infection
* With any other serious acute and chronic physical or mental disease or abnormal laboratory tests, which are likely to increase risks or interfere with the interpretation of the results, or researchers believe that patients are not suitable for enrollment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2013-01; Primary Completion 2018-12-30 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Overall survival | 5 years
  Overall survival is based on death from any cause, not just the condition being treated, thus it picks up death from side effects of the treatment, and effects on survival after relapse

SECONDARY OUTCOMES:
Treatment complication | 90 days
  defined as complications within the 90 days after treatment
Time to progress(TTP) | 3 years
  TTP: The Hazard Ratio will be analyzed respectively with 95% confidence interval. Meanwhile, Kaplan-Meier estimation and survival curves will be performed.
Disease control rate(DCR) | 3 years
  Disease control rate: Calculate the disease control rate of the two treatment groups (disease control rate) and its 95% confidence interval, and make a descriptive analysis.
Quality of life(Qol) | 5 years
  Quality of life: Follow the QOL-LC V2.0

CONTACTS AND LOCATIONS:
Overall Officials: Yunfei Yuan, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China